CLINICAL TRIAL: NCT02438865
Title: Prophylactic Intravesical Chemotherapy After Radical Nephroureterectomy for Upper Tract Urothelial Carcinoma: a Randomized Controlled Trial Between Single Postoperative Dose Versus Maintenance Therapy.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Magdy Elshabrawy, Fellow in Urology, Urology and Nephrology Center, Mansoura University, Mansoura, Egypt, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: MElsh112015
Record Dates: First submitted 2015-05-06; First posted 2015-05-08 (Estimated); Last update posted 2018-09-13 (Actual); Status verified 2018-09

CONDITIONS: Neoplasm, Ureter; Neoplasm, Bladder
Keywords: Upper Tract Urothelial Carcinoma; Intravesical Chemotherapy; Epirubicin; Urothelial Carcinoma
MeSH Terms: conditions — Ureteral Neoplasms; Urinary Bladder Neoplasms; Carcinoma, Transitional Cell

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Single instillation group (Active Comparator): will receive single intravesical dose of epirubicin intravesical therapy (50 mg) within 48 hours of radical nephroureterectomy with open bladder cuff excision.
  Interventions: Drug: Immediate instillation of intravesical chemotherapy-Epirubicin-
- Maintainance therapy group (Active Comparator): will receive a single intravesical dose of epirubicin and an additional 6 weekly doses of intravesical therapy (50 mg) after surgery then monthly maintenance therapy for 1 year.
  Interventions: Drug: Maintainance therapy of intravesical chemotherapy-Epirubicin-

INTERVENTIONS:
Drug: Immediate instillation of intravesical chemotherapy-Epirubicin-
  Arms: Single instillation group
Drug: Maintainance therapy of intravesical chemotherapy-Epirubicin-
  Arms: Maintainance therapy group

SUMMARY:
This clinical trial is designed to compare the effect of single postoperative intravesical chemotherapy instillation versus maintenance therapy on reducing bladder cancer recurrence after surgery for UTUC.

DETAILED DESCRIPTION:
INTRODUCTION Upper tact urothelial carcinoma (UTUC) arises from the urothelial lining of the urinary tract from the renal calyces to the ureteral orifice. It comprises 10 % of all renal tumors and 5% of all urothelial malignancies (Jemal et al., 2007). A common feature of UTUC is multiple anatomic locations in the urinary tract either synchronous or metachronous. While synchronous bladder tumor can be identified at time of evaluation of UTUC, recurrent bladder tumor remains a major concern.

Incidence of bladder recurrence after management of UTUC varies considerably from 20% - 50% (Kirkali and Tuzel., 2003; Hall et al., 1998). Although the risk factors for development of bladder tumor post surgical management of UTUC were previously studied, considerable variations were observed in the literature. In a recent meta-analysis, Seisen et al., in 2014 have identified male gender, previous bladder cancer, and preoperative chronic kidney disease as patient-specific predictors. While tumor-specific predictors were as follows: positive preoperative urinary cytology, ureteral location, multifocality, invasive stage, and necrosis. Lastly, treatment-specific predictors were a laparoscopic approach, extravesical bladder cuff removal, and positive surgical margins.

To date, two theories have been proposed for intravesical recurrence after radical nephroureterectomy including intraluminal seeding of a single transformed cell (Habuchi et al., 1993) and pan-urothelial field defect e.g. carcinogenic exposure of the entire urothelial tract can lead to independent multifocal development (Takahashi et al., 2001; Jones et al., 2005). Therefore, it has been suggested that administration of a single dose of intravesical chemotherapy in the early postoperative period might prevent seeding of transitional cancer cells and therefore might help reduce the incidence of urothelial tumor recurrence in the first year post surgery (O'Brien et al., 2011). To the best of our knowledge, only two randomized controlled trials have investigated this hypothesis (O'Brien et al., 2011; Ito et al., 2013 ). O' Brien et al., 2011, have reported 16% of patients in the mitomycin C arm and 27% of patients in the standard treatment arm developed bladder cancer recurrence within the first year postoperative. Ito et al., 2013, reported 16.9% of patients in the pirarubicin arm and 31.8% of patients in the standard treatment arm developed bladder cancer recurrence within the first postoperative year. Based on these findings, it has been recommended in the last European association of urology guidelines that postoperative instillation of chemotherapy is recommended to avoid bladder cancer recurrence "grade B recommendation" (Roupret et al., 2013).

In 2001 Sakamoto et al., examined the significance of intravesical instillation of Mitomycin C and cytosine arabinoside over 2 years period. They showed that instillation would reduce the recurrence rate in the bladder after surgery for upper urinary tract tumors. However, this study was underpowered to detect the desired difference. The investigators hypothesized that the 16% incidence of bladder tumor recurrence after single postoperative instillation of intravesical chemotherapy after surgery for UTUC might be attributed to the influence of pan-urothelial field defect theory. Therefore, the investigators assume that maintenance intravesical chemotherapy would significantly reduce this percentage of tumor recurrence.

AIM OF THE WORK This clinical trial is designed to compare the effect of single postoperative intravesical chemotherapy instillation versus maintenance therapy on reducing bladder cancer recurrence after surgery for UTUC.

PATIENTS AND METHODS

Patients:

Type of the study A randomized controlled trial (RCT), phase II.

Study locality Urology Nephrology Center (UNC)

Study design

Patients with UTUC will be prospectively randomized into two groups using excel software by random table function:

1. Group 1: will receive single intravesical dose of epirubicin intravesical therapy (50 mg) within 48 hours of radical nephroureterectomy with open bladder cuff excision.
2. Group 2: will receive a single intravesical dose of epirubicin and an additional 6 weekly doses of intravesical therapy (50 mg) after surgery then monthly maintenance therapy for 1 year.

Exclusion criteria

1. Patients with history of bladder tumor
2. Patients with synchronous bladder tumor
3. Patients with advanced stage (T4)

Power calculation and Statistical analysis All statistical analysis will be performed using IBM v. 20 statistical software and the statistical tests will be used appropriately whenever indicated. The calculation of sample size is conducted using G*power statistical software (Faul F et al., 2007). The recurrence rate in the control arm of the study was reported to be 16% after single intravesical dose of chemotherapy. If the expected treatment effect of maintenance chemotherapy was similar to that observed in bladder tumor, there would be a reduction in recurrence rate by 38% )Huncharek M et al., 2001). Therefore, to detect this level of difference at a power of 80% and 5% level of significance, 35 patients will be required to detect the difference between groups (1) and (2) and accounting for 15% losses in each arm, 40 patients will be randomized in each arm.

Methods:

Intervention Patients will be randomly allocated into one of the two groups using excel software by random table function at the day of surgery. Radical nephroureterectomy will be done through the open or laparoscopic approach while bladder cuff excision will be performed through the open approach. All data will be prospectively maintained and include patients' demographics, preoperative laboratory parameters, operative details and postoperative complications

Follow up The scheduled follow up will be according to the EUA guidelines (Roupret M et al., 2013) by scheduling a urine cytology and cystoscopy at 3 months then at one year while CT urography at one year for non-invasive tumors and at 6 months and one year for invasive tumors. All chemotherapy-related complications will be reported.

Outcome and end-point The primary outcome of the study is the diagnosis of intravesical recurrence within the first year after surgery. The secondary outcome is to determine the adverse events postoperative morbidity, mortality and survival of patients with UTUC.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with UTUC without history of bladder tumor
2. Patients with UTUC without synchronous bladder tumor

Exclusion Criteria:

1. Patients with history of bladder tumor
2. Patients with synchronous bladder tumor
3. Patients with advanced stage (T4)

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2018-05-01 (Actual); Study Completion 2018-05-30 (Actual)

PRIMARY OUTCOMES:
bladder recurrence | 1 year after surgery
  The primary outcome of the study is the diagnosis of intravesical recurrence within the first year after surgery.

SECONDARY OUTCOMES:
adverse events | 1 year after surgery
  The secondary outcome is to determine the adverse events postoperative morbidity, mortality and survival of patients with UTUC.

CONTACTS AND LOCATIONS:
Overall Officials: Yasser M. Osman, MD, Study Director — Urology And Nephrology Center, Mansoura University, Mansoura
Locations (1):
- Urology and Nephrology Center, Al Mansurah, DK, Egypt